CLINICAL TRIAL: NCT03559998
Title: Learning Process of Fourth Year Medical Students During an Obligatory Doctor-patient Relationship Training, Including Role Play, Simulated Consultation, Balint Group and Courses: a Mixed Method Study
Brief Title: Learning Process of Fourth Year Medical Students During a Doctor-patient Relationship Training
Acronym: APTHERA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation Friedlander (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI18026HLJ; 2018-A00385-50 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Undergraduate Medical Students' Learning Process in Doctor-patient Relationship Training
Keywords: Simulation training; role-play; psychiatry; students; medical; psychology; educational; learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: lecture — * Empathy (1 hour)
  * Doctor- patient relationship (1, 5 hour)
  Other Names: Empathy and doctor-patient relationship
Other: Simulation using Role play — * serious illness announcement
  * abuse demand management
  * reticent patient management
  Other Names: Doctor-patient relationship role play
Other: Discussion group — Share about clinical work experience and elaboration about psychoaffective and relational challenge
  Other Names: Balint Group
Other: Simulation using Simulated patient — * HIV announcement
  * Refuse of antibiotic prescription
  Other Names: Objective Structured Clinical Examination (OSCE)

SUMMARY:
This study aims to explore learning process for undergraduate students in this doctor-patient relationship course. This study is one of the 3 studies included in a PhD on learning process during simulation training in psychiatry. The results of this 3 studies will aim at building a formative and summative assessment tool of competences specific to this pedagogic context.

DETAILED DESCRIPTION:
Methodology: Mixed method study with:

Qualitative : Grounded Theory analysis of :

* Semi-structured interview of learners and teachers
* Learning written traces of students

Quantitative features:

* Self-reported questionnaires on satisfaction
* Sociodemographical data and others questions

ELIGIBILITY:
Inclusion Criteria:

* Age > to 18 years old
* Undergraduate medical fourth-year student of Paris Descartes University
* Taking part in an obligatory doctor-patient relationship training, including role play, simulated consultation, Balint group and courses
* Draw by lot
* French or English language
* Agreement

Exclusion Criteria:

* Refusal of agreement
* Undergraduate medical fourth-year student of Paris Descartes University who couldn't take part in an obligatory doctor-patient relationship training, including role play, simulated consultation, Balint group and courses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Undergraduate medical fourth-years student of Paris Descartes University. To diversify recruitment of students for semi-structured interview, investigators will conduct a drawing of lot, thanks to a computer programm, until data saturation.
  Apprenticeship trace will also be drawn of lot, until data saturation.
Sampling Method: Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2018-06-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Learning processes | 2 hours
  Learning processes according to students and teachers' perspective evaluated by face-to-face semi-structured interviews, faced with analysis of students' written apprenticeship traces

SECONDARY OUTCOMES:
supporting or preventing factors of learning | 2 hours
  according to students and teachers' perspective evaluated by face-to-face semi-structured interviews, faced with analysis of students' written apprenticeship traces

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Aude PIOT, MD, PhD, Principal Investigator — Paris Descartes University, France; Bruno FALISSART, MD, PhD, Study Chair — Paris Saclay South University, Faculty of medicine, Orsay, France; Antoine TESNIERE, Md, PhD, Study Chair — University of Paris 5 - Rene Descartes
Locations (1):
- Paris Descartes University, Sorbonne Paris City, Faculty of Medicine, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
For data about satisfaction and sociodemographic, it will be collected on a commun and secured base so as to support confrontation of analysis.
  For qualitative data, they will be kept on secured informatics interface (of Dr Marie-Aude Piot) of University Hospital Institute "Mutualiste Montsouris". The qualitative researchers will have access to this base for data quotation.
Supporting Information: Study Protocol
Time Frame: From data collection (june-july 2018 to data saturation estimated at December 2018)
Access Criteria: Only researchers involved in data analysis